CLINICAL TRIAL: NCT04298723
Title: Randomized Comparison of Interventional Closure of the Left Atrial Appendage Using a LAA Closure Device Versus Oral Anticoagulation Therapy in Patients With Non-valvular Atrial Fibrillation and Status Post Intracranial Bleeding.
Brief Title: Comparison of LAA-Closure vs Oral Anticoagulation in Patients With NVAF and Status Post Intracranial Bleeding.
Acronym: CLEARANCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: KCRI (Other)
Responsible Party: Principal Investigator, Sven Möbius-Winkler, Principal Investigator, Debuty director cardiology departement, Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZKSJ0123_Clearance
Record Dates: First submitted 2020-03-01; First posted 2020-03-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-02

CONDITIONS: Intracranial Hemorrhages; Atrial Fibrillation (AF); Atrial Flutter
Keywords: Intracranial Hemorrhage; Intracranial Bleeding; Atrial Fibrillation; Anticoagulation; LAA Occlusion
MeSH Terms: conditions — Intracranial Hemorrhages; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, randomized, controlled, non-blinded clinical trial with a two-arm parallel group design
Who Masked: Outcomes Assessor
Masking Description: CEC blinded DSMB blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left Atrial Appendage Occlusion (Experimental): Percutaneous closure of the LAA by use of CE-mark approved LAA occlusion device Watchman / Watchman FLX
  Interventions: Device: Percutaneous closure of the LAA (Watchman / Watchman FLX)
- Best Medical Therapy for Anticoagulation (No Intervention): Standard of care (according to current guidelines)

INTERVENTIONS:
Device: Percutaneous closure of the LAA (Watchman / Watchman FLX) — LAA closure procedure will be done by experienced operators according to the local SOP. LAA closure will be performed under fluoroscopic and TEE guidance within conscious sedation or general anesthesia. Antibiotic single-shot prophylaxis should be administered peri-procedurally (i.e., cefazolin 2 g). The specific anatomy of the LAA is evaluated and an appropriately sized CE-marked device (Watchman or Watchman FLX) is deployed. LAA angiography and TEE imaging is performed to identify optimal positioning of the device and to exclude a relevant leak. Following device deployment, patients will receive a therapy according to the manufacturers IFU, currently Aspirin and clopidogrel for 3 months followed by single Aspirin up to 12 months. Alternatively, 3 months of NOAC followed by Aspirin monotherapy up to 12 months are possible.
  Arms: Left Atrial Appendage Occlusion

SUMMARY:
Atrial fibrillation is the most common cardiac arrhythmia. In atrial fibrillation, there is a risk that clots can form in the heart, especially in the left atrium. If these clots come loose, there is a risk of stroke. To prevent strokes, patients with atrial fibrillation and status post ICB can be treated with anticoagulants. This medication therapy prevents blood clots from forming in the heart, but can also cause bleeding. Another therapy option is the occlusion of the left atrium. After closure of the left atrium, only a short anticoagulation therapy is necessary until the occluder has healed. The aim of the study is to compare these two treatment approaches. In this study only already approved drugs and occlusion systems will be used.

DETAILED DESCRIPTION:
Within the current trial, two novel strategies are tested in a randomized fashion in patients with atrial fibrillation and status post intracranial bleeding. Patients with ICH were usually excluded from the large NOAC trials and were also not representatively included in the large Watchman device trials. On the other hand, registries show that there is a significant proportion of patients with status post ICH that were implanted with a LAA closure device in clinical routine, and also there are those patients treated with NOAC due to their high stroke risk, despite the risk of recurrent ICH.

Both therapies, NOAC and LAA closure are effective in preventing stroke in patients with AF at high risk for stroke. Also, for both therapies there is evidence for prevention of bleedings, especially intracranial bleeding events.

Patients within the LAA closure group will have the chance after successful closure of the LAA to quit oral anticoagulation medication and therefore reduce their lifetime risk for bleeding and recurrent bleeding. Patients in the NOAC group are provided with an excellent protection against stroke and a significant reduced bleeding risk compared to Vitamin K antagonist therapy.

The trial will help to develop data and hopefully guidelines for management of patients with AF and status post intracranial bleedings. It may help to give physicians data to therapy patients post ICH adequately and help to reduce mortality rates in those patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Documented atrial fibrillation (paroxysmal, persistent, long-standing persistent or permanent)
* CHA2DS2VASc-Score ≥2
* Status post intracranial bleeding >6 weeks
* Favorable LAA anatomy
* Subject eligible for a LAA occluder device
* Age ≥18 years

Exclusion Criteria:

* Comorbidities other than AF requiring chronic (N)OAC therapy, e.g. mechanical heart valve prosthesis, hereditary thrombophilia requiring livelong OAC - recurrent thrombosis
* Symptomatic carotid disease (if not treated)
* Thrombus in the left atrium or left atrial appendage
* Active infection or active endocarditis or other infections resulting in bacteremia
* Functional Impairment (modified ranking scale ≥4 )
* Severe liver failure (Child-Pugh class C or liver failure with coagulopathy)
* Pregnancy or breastfeeding
* Subject with participation in another interventional clinical trial during this study or within 30 days before entry into this trial.
* Known terminating disease with life expectancy <1 year (including those with end-stage heart failure)
* Subjects, who are committed to an institution due to binding official or court order
* Subjects with planned cardiac or non-cardiac surgery or intervention. (These subjects can be included 30 days after intervention / surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Event free survival of the composite of cardiovascular or unexplained death, stroke (including ischemic or hemorrhagic stroke), systemic embolism, bleeding (BARC type 2-5) | up to 3 years after randomization
  Cardiovascular or unexplained death
  Cardiovascular mortality:
  * Death due to proximate cardiac cause e.g. myocardial infarction, cardiac tamponade, worsening heart failure, or endocarditis
  * Death caused by non-coronary, non-CNS vascular conditions such as: pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm or other vascular disease
  * Death from vascular CNS causes from hemorrhagic and ischemic stroke
  * All procedure-related deaths including those related to a complication of the procedure or treatment for a complication of the procedure
  * Sudden or unwitnessed death defined as non-traumatic, unexpected fatal event occurring within one hour of the onset of symptoms in an apparently healthy subject. If death is not witness, the definition applies when the victim was in good health 24 hours before the event
  * Death of unknown cause
Event free survival of the composite of cardiovascular or unexplained death, stroke (including ischemic or hemorrhagic stroke), systemic embolism, bleeding (BARC type 2-5) | up to 3 years after randomization
  Stroke (including ischemic or hemorrhagic stroke) - A stroke is an acute episode (lasting >24 hours) of focal neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction. Strokes are characterized as follows:
  * Ischemic stroke: an acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction of the central nervous system tissue. Hemorrhage may be a consequence of ischemic stroke. In this situation, the stroke is an ischemic stroke with hemorrhagic transformation and not a hemorrhagic stroke.
  * Hemorrhagic stroke: an acute episode of focal or global cerebral or spinal dysfunction caused by intraparenchymal, intraventricular, or subarachnoid hemorrhage
Event free survival of the composite of cardiovascular or unexplained death, stroke (including ischemic or hemorrhagic stroke), systemic embolism, bleeding (BARC type 2-5) | up to 3 years after randomization
  Systemic embolism - Non-CNS systemic embolism is defined as abrupt vascular insufficiency of an extremity or organ associated with clinical or radiological evidence of arterial occlusion in the absence of other likely mechanisms, (e.g., trauma, atherosclerosis, instrumentation). In the presence of atherosclerotic peripheral vascular disease, diagnosis of embolism to the lower extremities should be made with caution and requires angiographic demonstration of abrupt arterial occlusion.
Event free survival of the composite of cardiovascular or unexplained death, stroke (including ischemic or hemorrhagic stroke), systemic embolism, bleeding (BARC type 2-5) | up to 3 years after randomization
  Bleeding (BARC type 2-5) - Type 2
  Any clinically overt sign of hemorrhage that "is actionable" and requires diagnostic studies, hospitalization, or treatment by a health care professional
  Type 3
  1. Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed); transfusion with overt bleeding
  2. Overt bleeding plus hemoglobin drop < 5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents
  3. Intracranial hemorrhage confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision
  Type 4
  CABG-related bleeding within 48 hours
  Type 5
  1. Probable fatal bleeding
  2. Definite fatal bleeding (overt or autopsy or imaging confirmation)

SECONDARY OUTCOMES:
Cardiovascular or unexplained death per year; Stroke per year; Systemic embolism per year; Bleeding per Year | up to 3 years after randomization
  Primary endpoint events per year: Cardiovascular or unexplained death per year; Stroke per year; Systemic embolism per year; Bleeding per Year; The study participants or, if consent has been obtained, relatives are questioned during the visits, if necessary, diagnostic results are obtained;
Combined endpoint: MACCE | up to 3 years after randomization
  Combined endpoint: MACCE (stroke/systemic embolism/cardiovascular death/myocardial infarction)
Mortality | up to 3 years after randomization
  Mortality (including all-cause death, cardiovascular death, non- cardiovascular
Bleeding (BARC type 2-5) | up to 3 years after randomization
  Type 2
  Any clinically overt sign of hemorrhage that "is actionable" and requires diagnostic studies, hospitalization, or treatment by a health care professional
  Type 3
  1. Overt bleeding plus hemoglobin drop of 3 to < 5 g/dL (provided hemoglobin drop is related to bleed); transfusion with overt bleeding
  2. Overt bleeding plus hemoglobin drop < 5 g/dL (provided hemoglobin drop is related to bleed); cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring IV vasoactive agents
  3. Intracranial hemorrhage confirmed by autopsy, imaging, or lumbar puncture; intraocular bleed compromising vision
  Type 4
  CABG-related bleeding within 48 hours
  Type 5
  1. Probable fatal bleeding
  2. Definite fatal bleeding (overt or autopsy or imaging confirmation)
Systemic embolism | up to 3 years after randomization
  Non-CNS systemic embolism is defined as abrupt vascular insufficiency of an extremity or organ associated with clinical or radiological evidence of arterial occlusion in the absence of other likely mechanisms, (e.g., trauma, atherosclerosis, instrumentation). In the presence of atherosclerotic peripheral vascular disease, diagnosis of embolism to the lower extremities should be made with caution and requires angiographic demonstration of abrupt arterial occlusion.
Ischemic stroke | up to 3 years after randomization
  An acute episode of focal cerebral, spinal, or retinal dysfunction caused by infarction of the central nervous system tissue. Hemorrhage may be a consequence of ischemic stroke. In this situation, the stroke is an ischemic stroke with hemorrhagic transformation and not a hemorrhagic stroke.
Hemorrhagic stroke | up to 3 years after randomization
  An acute episode of focal or global cerebral or spinal dysfunction caused by intraparenchymal, intraventricular, or subarachnoid hemorrhage
Myocardial infarction | up to 3 years after randomization
  A detailed description of the criteria for myocardial infarction can be found in the study protocol.
Hospitalization for bleeding or cardiovascular event | up to 3 years after randomization
  Hospitalization for bleeding or cardiovascular event
Intracranial bleeding | up to 3 years after randomization
  Intracranial bleeding

OTHER OUTCOMES:
Secondary Safety Endpoints | As indicated within description.
  * Periprocedural complications within 7 days combined from: pericardial effusion, stroke, major bleeding, device embolization, intracranial bleeding, air embolism
  * Device related thrombus/fracture/erosion
  * Vascular access related complications requiring intervention
  * Procedure-related death
  * Technical and procedural success of device implantation (LAA closure)
  * Post-procedure infection rate
  * Periprocedural outcomes at 7 and 45 calendar days after implantation
  * Bleeding requiring transfusion (BARC 2-5)
  * Air embolism

CONTACTS AND LOCATIONS:
Overall Officials: Sven Möbius-Winkler, Prof. Dr., Principal Investigator — Department of Internal Medicine I, Jena University Hospital; Albrecht Günther, Dr., Principal Investigator — Department of Neurology, Jena University Hospital; Christian Senft, Prof. Dr., Principal Investigator — Department of Neurosurgery, Jena University Hospital; P. Christian Schulze, Prof. Dr., Principal Investigator — Department of Internal Medicine I, Jena University Hospital
Locations (33):
- Germany (30):
  - University Hospital Mannheim, Mannheim, Baden-Wurttemberg
  - RHÖN-KLINIKUM Campus Bad Neustadt, Bad Neustadt an der Saale, Bavaria
  - Therapiezentrum Burgau, Burgau, Bavaria
  - REGIOMED Klinikum Coburg, Coburg, Bavaria
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum Ingolstadt, Ingolstadt, Bavaria
  - RoMed Klinikum, Rosenheim, Bavaria
  - Cardiologicum Hamburg, Hamburg, Hamburg
  - Asklepios Klinik Wandsbek, Hamburg, Hamburg
  - Asklepios Klinik Nord Heidberg, Hamburg, Hamburg
  - Asklepios Klinik Altona, Hamburg, Hamburg
  - Herz-Kreislauf-Zentrum, Rotenburg an der Fulda, Hesse
  - Evangelisches Klinikum Bethel, Bielefeld, North Rhine-Westphalia
  - Klinikum Dortmund, Dortmund, North Rhine-Westphalia
  - Knappschaft Kliniken, Dortmund, North Rhine-Westphalia
  - Westpfalz-Klinikum, Kaiserslautern, Rhineland-Palatinate
  - Katholisches Klinikum Koblenz • Montabaur, Koblenz, Rhineland-Palatinate
  - Klinikum Chemnitz, Chemnitz, Saxony
  - Dresden Heart Center, Dresden, Saxony
  - University Hospital Leipzig, Leipzig, Saxony
  - Klinikum St. Georg, Leipzig, Saxony
  - Heart Center Leipzig, Leipzig, Saxony
  - Helios Klinikum Pirna, Pirna, Saxony
  - Heinrich-Braun-Klinikum (HBK), Zwickau, Saxony
  - University Hospital Magdeburg, Magdeburg, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein (UKSH), Lübeck, Schleswig-Holstein
  - Charité - Universitätsmedizin Berlin (CBF), Berlin, State of Berlin
  - Charité - Universitätsmedizin Berlin (CVK, Berlin, State of Berlin
  - Helios Klinikum Erfurt, Erfurt, Thuringia
  - University Hospital Jena, Jena, Thuringia
- Poland (3):
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan, Greater Poland Voivodeship
  - Polsko-Amerykańskie Kliniki Serca, Bielsko-Biala, Silesian Voivodeship
  - Górnośląskim Centrum Medycznym, Katowice, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No